CLINICAL TRIAL: NCT02935816
Title: Whole Body Multi---Parametric MRI: Accuracy in Staging of Biochemically Relapsed Prostate Cancer
Brief Title: Localising Occult Prostate Cancer Metastases With Advanced Imaging TEchniques
Acronym: LOCATE
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University College, London (Other)
Responsible Party: Sponsor
Other Study IDs: 15/0047
Record Dates: First submitted 2015-12-01; First posted 2016-10-18 (Estimated); Last update posted 2016-10-18 (Estimated); Status verified 2015-12

CONDITIONS: Prostate Cancer
MeSH Terms: conditions — Prostatic Neoplasms

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — 100 ml of blood sample for exosome analysis
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Radiation: Whole body MRI — We have developed and assessed the feasibility of performing whole---body multi---parametric MRI for staging metastatic disease. We hypothesize that a whole body multi---parametric MRI will be more sensitive and specific than conventional imaging staging for detection of metastatic disease in patients with biochemical failure following local therapies. We therefore propose a comparative trial of conventional imaging verses whole---body multi---parametric MRI within this population of men

SUMMARY:
The investigator prospectively compare diagnostic concordance of whole body multi---parametric Magnetic Resonance Imaging (MRI) with current conventional multi---modality reference standard imaging (CT scan, isotope bone scan +/--- PET---CT scan) for staging of prostate cancer patients with biochemical relapse following external beam radiotherapy or brachytherapy of locally advanced prostate cancer.

DETAILED DESCRIPTION:
The investigators have developed and assessed the feasibility of performing whole---body multi---parametric MRI for staging metastatic disease. The investigators hypothesize that a whole body multi---parametric MRI will be more sensitive and specific than conventional imaging staging for detection of metastatic disease in patients with biochemical failure following local therapies. Investigators therefore propose a comparative trial of conventional imaging verses whole---body multi---parametric MRI within this population of men. The investigators would further like to explore whether heterogeneity between metastases of multi---parametric MRI signals can predict men unlikely to respond to ADT. The investigators aim to enhance the main study by exploratory work on exosome, pathway and genomic analysis, the results of which could lead to complimentary imaging / non---imaging biomarker combinations of clinical utility for patient stratification. Finally the investigators will perform a health economic analysis to assess the cost---effectiveness of whole---body multi---parametric MRI for metastatic disease staging compared with conventional staging with computed tomography and bone---scans.

ELIGIBILITY:
Inclusion Criteria:

* Men who have undergone previous external beam radiotherapy or brachytherapy with or without neo---adjuvant/adjuvant hormone therapy
* Men who have radiorecurrent disease defined by biochemical failure - Phoenix definition (PSA nadir + 2 ng/mL)

Exclusion Criteria:

* Men unable to have MRI scan, or in whom artefact would significantly reduce quality of MRI
* Men unable to give informed consent

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Prostaete cancer patients with biochemical relapse following external beam radiotherapy or brachytherapy of locally advanced prostate cancer.
Sampling Method: Non-Probability Sample
Enrollment: 130 (Estimated)
Dates: Start 2015-01; Primary Completion 2018-01 (Estimated); Study Completion 2018-01 (Estimated)

PRIMARY OUTCOMES:
The investigator will measure and analyse sensitivity and specificity of WB-MRI compared to conventional multi-modality imaging for detection of regional lymph node distant metastasis.T | 3 years

SECONDARY OUTCOMES:
Interobserver agreement for WB-MRI: Per-site and per-nodal staging assessment will be done by two radiologists separately and then in consensus. Kappa agreement statistic will be tested for the level of agreement for per-site and per-patient assessments. | 3 years
The investigator will investigate whether there would be any significant correlation between MRI quantitative parameters and the response following treatment. | 3 years
The investigator will evaluate using blood test differences between two groups | 3 years
  The investigator will evaluate using blood test, differences between Human Epidermal growth factor Receptor analysis in patients with castrate-resistant metastatic prostate cancer and non-metastatic patient to explore any significant differences between two groups
The investigator will asses the Cost-effectiveness by comparing the direct and indirect costs of multi-modality imaging path versus WB-MRI path | 3 years
The investagator will measure sensitivity and specificity of WB-MRI compared to choline PET-CT for detection of regional lymph node distant metastasis. Analysis of sensitivity and specificity will be investigated on per-site basis and per-patient basis | 3 years

CONTACTS AND LOCATIONS:
Overall Officials: Shonit Punwani, Principal Investigator — Centre for Medical Imaging
Locations (1):
- Centre for Medical Imaging, London, United Kingdom

IPD SHARING:
Plan to Share IPD: Yes

REFERENCES:
- [Derived] Adeleke S, Latifoltojar A, Sidhu H, Galazi M, Shah TT, Clemente J, Davda R, Payne HA, Chouhan MD, Lioumi M, Chua S, Freeman A, Rodriguez-Justo M, Coolen A, Vadgama S, Morris S, Cook GJ, Bomanji J, Arya M, Chowdhury S, Wan S, Haroon A, Ng T, Ahmed HU, Punwani S. Localising occult prostate cancer metastasis with advanced imaging techniques (LOCATE trial): a prospective cohort, observational diagnostic accuracy trial investigating whole-body magnetic resonance imaging in radio-recurrent prostate cancer. BMC Med Imaging. 2019 Nov 15;19(1):90. doi: 10.1186/s12880-019-0380-y. PMID 31730466